CLINICAL TRIAL: NCT02959359
Title: The Role of DAA in Reducing the Risk of Recurrence After Curative Treatment of HCC in Patients With Chronic Hepatitis C and Early Stage HCC
Brief Title: DAA in the Risk of Recurrence After Curative Treatment of HCC
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The supplies of study drug were halted by Gilead Sciences Ltd.
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); China Medical University Hospital (Other); Chi Mei Medical Hospital (Other); Chiayi Christian Hospital (Other); National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other); Tri-Service General Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, vghtpe user, Professor Yi-Hsiang Huang, Taipei Veterans General Hospital, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GILEAD IN-US-337-4109
Record Dates: First submitted 2016-10-30; First posted 2016-11-09 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Chronic hepatitis C; Hepatocellular Carcinoma; Direct-acting antiviral (DAA); Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C, Chronic; Recurrence | interventions — ledipasvir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DAA treatment arm (Other): Active DAA treatment ('Ledipasvir 90mg/Sofosbuvir 400 mg plus Ribavirin' ) for HCV-HCC patients after curative resection or ablation.
  Interventions: Drug: Ledipasvir 90mg/Sofosbuvir 400 mg; Drug: Ribavirin

INTERVENTIONS:
Drug: Ledipasvir 90mg/Sofosbuvir 400 mg — A 12 week Harvoni (Ledipasvir 90mg/Sofosbuvir 400 mg ) plus ribavirin will be provided after confirmation of curative treatment.
  Other Names: DAA
Drug: Ribavirin — A 12 week Harvoni (Ledipasvir 90mg/Sofosbuvir 400 mg ) plus ribavirin will be provided after confirmation of curative treatment.
  Other Names: rebetol

SUMMARY:
For early stage of HCC, surgical resection or radiofrequency ablation (RFA) is the mainstay curative treatments. However, recurrence is still a major issue after the surgery or RFA. Only selected patients are eligible and tolerable to IFN-based treatment after surgical resection and the sustained virological response varied.

Harvoni for genotype 1 HCV and sovaldi plus ribavirin for genotype 2 HCV can achieve high SVR and being recommended by AASLD and EASL. Mixed HCV genotype infection accounts for 10% of CHC patients in Taiwan. Sovaldi-based treatment plus ribavirin should be as effective as Sovaldi plus rivavirin in the treatment of genotype 2 HCV, as well as mixed genotype 1 and 2 HCV infection. As genotype 1 and 2 are the leading HCV genotypes in Taiwan, It can simplify the regimen of anti-HCV treatment in Taiwan by using Harvoni plus ribavirin, not only for genotype 1 and 2 HCV but also for mixed genotype 1 and 2 HCV infection. Although an unexpected high recurrence rate in HCC patients under DAA treatment was reported once. However, one recent study showed a low risk of HCC recurrence after DAA treatment. In this study, the investigators plan to enroll 130 HCV-HCC patients after confirming curative treatment for their HCC, either by surgery or RFA. For the cases fulfilling the inclusion/exclusion criteria, a 12 weeks Harvoni plus ribavirin treatment will be provided for all cases (single armed design). The primary objective of the study is annual recurrence-free survival after curative resection of HCV-HCC for up to 5 years. A hospital-based cohorts of HCV-related HCC undergoing surgical resection or RFA from Taipei Veterans General Hospital and Investigated Sites will be recruited as historical controls.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is a major etiology of hepatocellular carcinoma (HCC). For early stage of HCC, surgical resection or radiofrequency ablation (RFA) is the mainstay curative treatments. However, recurrence is still a major issue after the surgery or RFA. According to our previous report, the cumulated recurrence rate for small HCV-HCC was 72.4% at 5 year. PEG-interferon plus RBV treatment is the standard of care for chronic hepatitis C (CHC) in Taiwan. NHIRD data showed that PEG-IFN plus RBV treatment can reduce 12% of recurrence rate in 5 years (64% vs 52%) after curative resection of HCC. However, only selected patients are eligible and tolerable to IFN-based treatment after surgical resection and the sustained virological response varied.

Harvoni for genotype 1 HCV and sovaldi plus ribavirin for genotype 2 HCV can achieve high SVR and being recommended by AASLD and EASL. All-oral regimen, being more tolerable and effective for HCC patients after curative treatment than IFN-based treatment. Mixed HCV genotype infection accounts for 10% of CHC patients in Taiwan. Sovaldi-based treatment plus ribavirin should be as effective as Sovaldi plus rivavirin in the treatment of genotype 2 HCV, as well as mixed genotype 1 and 2 HCV infection. As genotype 1 and 2 are the leading HCV genotypes in Taiwan, It can simplify the regimen of anti-HCV treatment in Taiwan by using Harvoni plus ribavirin, not only for genotype 1 and 2 HCV but also for mixed genotype 1 and 2 HCV infection. Although an unexpected high recurrence rate in HCC patients under DAA treatment was reported once. However, one recent study showed a low risk of HCC recurrence after DAA treatment. Harvoni is an all-oral regimen, being more tolerable and effective for HCC patients after surgery than IFN-based treatment. The all oral regimen would be beneficial in eradicating HCV viral load and subsequently reduce the risk of recurrence after curative resection of HCV-HCC.

In this study, the investigators plan to enroll 130 HCV-HCC patients after confirming curative treatment for their HCC, either by surgery or RFA. For the cases fulfilling the inclusion/exclusion criteria, a 12 weeks Harvoni plus ribavirin treatment will be provided for all cases (single armed design). The primary objective of the study is annual recurrence-free survival after curative resection of HCV-HCC for up to 5 years. The secondary objectives of the study are SVR 4/12/24 by DAA, regression of fibrosis, incidence of liver-related complications (EV bleeding, ascites) after DAA treatment, and overall survival for 5 years.

A hospital-based cohorts of HCV-related HCC undergoing surgical resection or RFA from Taipei Veterans General Hospital and Investigated Sites will be recruited as historical controls. The historical controls include HCV-HCC undergoing curative treatment without Peg-interferon plus ribavirin treatment (cohort 1) or with Peg-interferon plus ribavirin treatment (cohort 2) after curative treatment (surgical resection or RFA) for HCC.

ELIGIBILITY:
Inclusion Criteria:

* Anti-HCV positive and HBsAg-negative
* HCV genotype 1 or 2 infection, mixed infection GT 1 & 2 is allowed
* HCV RNA ≥ 10,000 IU/ml at the time of screening
* Age > 20 y/o
* BCLC stage 0 or A HCC confirmed by pathology and receiving the first time of curative treatment
* No recurrence of HCC confirmed by contrast-enhanced image studies (CT or MRI) within 3 months post the curative treatment.
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-1
* Child-Pugh score ≤7

Exclusion Criteria:

* HBV, or HIV coinfection
* Co-existing other malignancy
* Intolerance to ribavirin
* Marked decompensated liver cirrhosis (CTP score>7)
* Uremia or renal impaired patients (eGFR<30)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is annual recurrence-free survival after curative resection of HCV-HCC for up to 5 years. | up to 5 years
  The primary objective of the study is annual recurrence-free survival after curative resection of HCV-HCC for up to 5 years.

SECONDARY OUTCOMES:
SVR 4/12/24 by DAA | up to 5 years
  SVR: sustained virological response. DAA: direct antiviral agent. SVR 4/12/24 means undetectable HCV viral load 4/12/24 weeks after completing DAA treatment.
Regression of fibrosis | up to 5 years
  Regression of fibrosis
Incidence of liver-related complications (EV bleeding, ascites) after DAA treatment | up to 5 years
  Incidence of liver-related complications (EV bleeding, ascites) after DAA treatment
Overall survival | up to 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsiang Huang, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided